CLINICAL TRIAL: NCT04518176
Title: Clinical Outcomes of Bilateral Uterine Artery Ligation During the Cesarean Delivery of Twins: A Randomized Controlled Trial
Brief Title: Bilateral Uterine Artery Ligation During the Cesarean Delivery of Twins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/279/8/18
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Masking Description: open label randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients with twin pregnancy undergoing cesarean section underwent bilateral uterine artery ligation and received oxytocin.
  Interventions: Procedure: bilateral uterine artery ligation; Drug: Oxytocin
- control group (Active Comparator): patients with twin pregnancy undergoing cesarean section received oxytocin only.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Procedure: bilateral uterine artery ligation — The peritoneum over the vesico-uterine pouch already being incised horizontally, the peritoneum over the uterine isthmus and cervix was dissected downwards, and this dissection was then extended laterally
  Other Names: BUAL
  Arms: study group
Drug: Oxytocin — 20 units by slow intravenous drip injection

SUMMARY:
Objective to assess the effectiveness of prophylactic bilateral uterine artery ligation (BUAL) in reducing the incidence of postpartum hemorrhage during cesarean delivery among women with twin pregnancy

DETAILED DESCRIPTION:
A randomized clinical trial at Aswan University Maternity Hospital, Egypt. Women with twin pregnancy undergoing scheduled or emergency cesarean were randomized into two groups. In the BUAL group, women underwent BUAL before placental delivery; in the control group, women had cesarean delivery without BUAL. The primary outcome was the estimated blood loss during a cesarean

ELIGIBILITY:
Inclusion Criteria:

* women undergoing cesarean section
* twin pregnancy

Exclusion Criteria:

* Placenta previa.
* Ante-partum hemorrhage.
* patient refuse to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with twin pregnancy undergoing cesarean section
Enrollment: 400 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
mean Blood loss after placental separation | 30 minutes
  by using weight of soaked towels (weight of soaked towel - weight of dry towel) and amount of blood in suction set

SECONDARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 12 hours
  number pf participants with blood loss > 1000ml
The number of participant needed for blood transfusion | 24 hours
  Calculation of the number of participant needed for blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No